CLINICAL TRIAL: NCT01248117
Title: Investigator Sponsored Trial of Polypoidal Choroidal Vasculopathy (PCV) Evaluation Assessing High-Dose Ranibizumab (2.0mg) Prospectively
Brief Title: Safety Study of High-Dose Ranibizumab for Polypoidal Choroidal Vasculopathy
Acronym: PEARL2
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Retina Consultants of Hawaii (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Gregg T. Kokame / Managing Partner, Retina Consultants of Hawaii
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVF4929s
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Polypoidal Choroidal Vasculopathy
Keywords: PCV; polypoidal; choroidal; vasculopathy
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy; Vascular Diseases | interventions — Ranibizumab

ARMS (2):
- Previously Treated (Experimental): With prior anti-vegf therapy, only, no sooner than 30 days prior to enrollment into trial
  Interventions: Drug: ranibizumab 2.0mg
- Treatment-Naive (Experimental): Treatment-Naive: no previous treatment for PCV
  Interventions: Drug: ranibizumab 2.0mg

INTERVENTIONS:
Drug: ranibizumab 2.0mg — Monthly, intravitreal injection 0.05ml

SUMMARY:
Monthly, continuous anti-vegf therapy for patients presenting with active polypoidal choroidal vasculopathy. Two arms, treatment naive and previously treated with an FDA approved anti-VEGF therapy, will be randomized and dosed with open label 2.0mg ranibizumab.

DETAILED DESCRIPTION:
Patients will be followed with spectral oct, 4m BCVA, ICG, FA and monthly eye examinations for one year.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age >= 25 years
* Polypoidal choroidal vasculopathy as noted on fluorescein and ICG angiography: active leakage, active bleeding or recent decrease in vision
* BVCA using ETDRS of 20/32 to 20/400

Exclusion Criteria:

* Any history of prior vitrectomy
* Any prior treatment with verteporfin PDT in the study eye
* Previous cataract surgery within the preceding 2 months of D0
* Active intraocular inflammation in the study eye
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* A condition, that in the opinion of the investigator, would preclude participation in the study (e.g. unstable medical status including blood pressure, cardiovascular disease)
* Participation in another investigational trial within 30 days of randomization that involved treatment with any drug that has not received regulatory approval at the time of study entry.
* Prior anti-VEGF (Macugen, Avastin, Lucentis) in the study eye within 30 days prior to enrollment in this study
* Known allergy to any component in the study drug
* Uncontrolled hypertension: >180/110
* major surgery within 28 days prior to randomization
* Myocardial infarction, other cardia events requiring hospitalization within 6 months prior to randomization
* Systemic anti-VEGF or pro-VEGF within 3 months of randomization
* Pregnancy or lactation
* History of recurrent significant infections or bacterial infections

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-12 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of intravitreal injections of 2.0mg ranibizumab administered monthly in preventing vision loss | 1 year
  To evaluate the efficacy of intravitreal injections of 2.0mg ranibizumab administered monthly in preventing vision loss, as measured by calculating the mean change in VA from baseline to Month 12

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of intravitreal injections of 2.0mg ranibizumab administered monthly | 1 year
  To evaluate the safety and tolerability of intravitreal injections of 2.0mg ranibizumab administered monthly
To evaluate the efficacy of monthly intravitreal injections of 2.0mg ranibizumab in preventing vision loss | 1 year
  To evaluate the efficacy of monthly intravitreal injections of 2.0mg ranibizumab in preventing vision loss as measured by the following: mean change from baseline in VA at 6 and 12 months, and the proportion of subjects who lose less than 5 letters of vision at Month 6 and Month 12.
To investigate the efficacy of monthly intravitreal injections of 2.0mg ranibizumab on clinical findings associated with PCV | 1 year
  the mean change from baseline at M6 to M12 of subretinal hemorrhage and/or exudates via fundus photographs and fundus exams, decrease and/or complete resolution of branching vascular network from PCV at M3, M6, and M12 as assessed by FA and ICG, decrease and/or complete resolution of the branching vascular network (BVN) from PCV at M3, M6, and M12, as assessed by FA and ICG, mean change in central foveal thickness and/or peripapillary edema as measured by SD-OCT in central and/or paracentral fields from baseline, M3, M6 and M12, incidence of ocular AEs

CONTACTS AND LOCATIONS:
Overall Officials: Gregg T Kokame, MD, MMM, Principal Investigator — Retina Consultants of Hawaii
Locations (2):
- United States (2):
  - Retina Consultants of Hawaii, Inc, Honolulu, Hawaii
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii